CLINICAL TRIAL: NCT01555177
Title: OCT Plaque and Thrombus IMaging in Patients Who Underwent Non-cardiac Surgery
Brief Title: Study of Coronary Plaque Rupture in Heart Attack Following Surgery Using Optical Coherence Tomography (OCT)
Acronym: OPTIMUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Victar Hsieh (Other)
Responsible Party: Sponsor-Investigator, Victar Hsieh, Interventional fellow, Hamilton Health Sciences Corporation
Organization: Hamilton Health Sciences Corporation (Other)
Other Study IDs: 12-099
Record Dates: First submitted 2012-03-09; First posted 2012-03-15 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Peri-operative Myocardial Infarction; Non-ST Elevation Myocardial Infarction
Keywords: Peri-operative myocardial infarction; Non-ST elevation myocardial infarction; Optical coherence tomography
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Peri-operative NSTEMI patients: Patients with POMI undergoing cardiac catheterization within 72 hours of first troponin elevation and within 2 weeks of their non-cardiac surgery.
- Non-surgery related NSTEMI patients: Patients with NSTEMI undergoing cardiac catheterization within 72 hours of symptom onset.

SUMMARY:
Background

It is commonly believed that a heart attack is caused by rupture of a plaque in the wall of the coronary artery, resulting in blood clots which impede blood flow. Currently, the investigators do not know whether heart attacks in patients who had a recent surgery are caused by the same disease process as those who did not have any surgery. This study will inform the investigators of very vital information about the cause of surgery-related heart attacks by taking images of coronary arteries using Optical Coherence Tomography (OCT). Images will also be taken from heart attack patients who did not have recent surgery, and the two groups will be compared.

OCT imaging

OCT is a relatively new imaging technology which is much better at taking images of the inside of the artery. OCT imaging procedure is carried out at the time of scheduled coronary angiogram, where a catheter with a mini-camera at its tip is advanced into the coronary artery, it will record video images of a length of the artery. These images will take approximately 3-4 seconds to obtain. Besides the OCT imaging being performed, the rest of the angiogram procedure is carried out in exactly the same way as it would normally proceed.

The OCT study will provide doctors with new information about the cause of surgery-related heart attacks, and will guide doctors in treating and preventing heart attacks in patients who undergo surgery.

Hypothesis

The investigators hypothesize that features of acute plaque rupture will be more common in patients with non-surgery related heart attacks compared to those which occur following surgery.

Design

Two groups of patients will be recruited(>20 in each group):

1. non-surgery related heart attack patients
2. patients who suffered from a heart attack following an operation.

Outcome measures

Using OCT, plaque features in coronary arteries of patients with heart attacks from both the surgical and non-surgical groups at the time of coronary angiogram will be compared.

DETAILED DESCRIPTION:
The majority of spontaneous non-ST segment elevation myocardial infarctions (NSTEMI) are attributed to rupture of an unstable atherosclerotic plaque in an epicardial coronary artery with thrombus formation. On the other hand, the pathophysiology underlying myocardial infarction following non-cardiac surgery is not well understood. The literature suggests that a significant proportion of myocardial infarctions following surgery may result from decreased myocardial perfusion in the presence of stable coronary artery disease without plaque rupture or thrombus formation.

Intra-coronary Optical Coherence Tomography (OCT) provides superior visualisation of the vascular lumen and structures close to the arterial lumen compared to IVUS, including features of plaque instability, including atherosclerotic plaque contents, fibrous cap thickness, thin cap fibroatheromas (TCFA), macrophage infiltration and calcium (2-10). OCT is therefore an ideal imaging technique to examine the pathophysiology involved in POMI, where features of plaque rupture and thrombus formation can be clearly distinguished from stable plaques.

An improved understanding of the pathophysiology of MI following non-cardiac surgery will guide management more appropriately.

Primary objective

1. To identify features of acute plaque rupture in peri-operative myocardial infarction (POMI)
2. To compare frequency of acute plaque rupture imaging findings between POMI and non-operative non-ST-elevation myocardial infarction (NSTEMI)

Hypothesis

The investigators hypothesize that features of acute plaque rupture will be more common in patients with non-operative NSTEMI compared to POMI.

Outcome measures

1. OCT features of coronary plaque rupture will be obtained at the time of coronary angiography, these features include thin cap fibroatheroma, intramural thrombus and plaque fissuring. OCT data from NSTEMI and POMI patient groups will be compared. Data on other plaque features, including fibrous cap thickness, lipid core, minimum luminal cross-sectional area (CSA), ruptured cavity CSA will also be collected, and compared between the two patient groups.

There will be no clinical follow-up in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Referred to coronary angiography with the view of revascularisation

Exclusion Criteria:

* ST elevation myocardial infarction
* Shock defined as the systolic blood pressure <90mmHg and tachycardia with heart rate >100 with evidence of systemic organ hypoperfusion.
* Inability to give consent
* Previous coronary artery bypass surgery due to the limited anticipated feasibility of OCT imaging in native vessels of patients with prior bypass grafts.
* PCI with stenting in the previous 6 months due to the elevated risk of stent related complications (thrombosis or restenosis) as the potential cause of the NSTEMI.
* GFR <35 due to need for additional 40-60 cc contrast during OCT imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSTEMI and peri-operative MI patients will be screened in the catheterisation laboratory. In addition, peri-operative MI patients will be screened in hospital wards, where patient referral for cardiac catheterisation will be based on clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Evidence of plaque rupture by OCT imaging | Day 1
  OCT evidence of plaque rupture, presence of white or red thrombus will be collected at the time of coronary angiography.

SECONDARY OUTCOMES:
Other features OCT features of atherosclerotic plaques. | Day 1
  lFeatures of stable plaques in the coronary artery, including: Lipid core, fibrous cap, thin cap fibroatheroma, thick cap fibroatheroma, minimum luminal cross-sectional area, ruptured cavity CSA.

CONTACTS AND LOCATIONS:
Overall Officials: Victar Hsieh, MBBS PhD, Principal Investigator — Hamilton Health Services; Tej Sheth, BArts SC MD, Principal Investigator — Hamilton Health Services
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada